CLINICAL TRIAL: NCT00064220
Title: A Phase II Study of Intravenous TZT-1027, Administered Weekly Times Two, Every Three Weeks, to Patients With Advanced or Metastatic Soft Tissue Sarcomas (STS) With Prior Exposure to Anthracycline-Based Chemotherapy
Brief Title: Soblidotin in Treating Patients With Advanced or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000310138; DAIICHI-1027A-PRT007; CPMC-IRB-20030512; MSKCC-03061
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Sarcoma
Keywords: adult leiomyosarcoma; adult malignant fibrous histiocytoma; adult liposarcoma; adult rhabdomyosarcoma; adult synovial sarcoma; adult fibrosarcoma; adult angiosarcoma; adult malignant hemangiopericytoma; stage IV adult soft tissue sarcoma; recurrent adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Leiomyosarcoma; Histiocytoma, Malignant Fibrous; Liposarcoma; Rhabdomyosarcoma; Sarcoma, Synovial; Fibrosarcoma; Hemangiosarcoma; Hemangiopericytoma, Malignant | interventions — soblidotin

INTERVENTIONS:
Drug: soblidotin

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as soblidotin use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of soblidotin in treating patients who have advanced or metastatic soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective tumor response rate in patients with advanced or metastatic soft tissue sarcoma with prior exposure to anthracycline-based chemotherapy when treated with soblidotin.
* Determine the duration of response in patients treated with this drug.
* Determine the time to tumor progression in patients treated with this drug.
* Determine the median survival time and 12-month survival rate of patients treated with this drug.
* Determine the quantitative and qualitative toxic effects of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive soblidotin IV over 1 hour on days 1 and 8. Treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for survival.

PROJECTED ACCRUAL: A total of 27 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed soft tissue sarcoma of 1 of the following tumor types:

  * Malignant fibrous histiocytoma
  * Liposarcoma
  * Rhabdomyosarcoma
  * Synovial sarcoma
  * Malignant paraganglioma
  * Fibrosarcoma
  * Leiomyosarcoma
  * Angiosarcoma, including hemangiopericytoma
  * Malignant peripheral nerve sheath tumor
  * Unclassified sarcoma
  * Miscellaneous sarcoma, including mixed mesodermal tumors of the uterus
* The following tumor types are not eligible:

  * Gastrointestinal stromal tumor
  * Chondrosarcoma
  * Malignant mesothelioma
  * Neuroblastoma
  * Osteosarcoma
  * Ewing's sarcoma
  * Embryonal rhabdomyosarcoma
* Evidence of disease progression
* Must have received 1 prior anthracycline-based chemotherapy regimen for metastatic disease

  * Adjuvant chemotherapy is not considered 1 prior regimen unless tumor progressed within 12 months of therapy
* At least 1 measurable lesion with indicator lesions outside of any prior radiation field
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age

* 15 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* SGOT and/or SGPT no greater than 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Bilirubin no greater than 1.5 times ULN

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* Ejection fraction at least 40% by MUGA

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No baseline neurotoxicity grade 2 or greater
* No concurrent serious infection
* No psychiatric disorder that would preclude giving informed consent or complying with study requirements
* No other concurrent severe or uncontrolled medical illness that would preclude study participation
* No other malignancy except nonmelanoma skin cancer, carcinoma in situ of the cervix, or any other malignancy for which the patient has been in complete remission and off all therapy for at least 5 years

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent anticancer biologic therapy

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy and recovered
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* Recovered from prior radiotherapy
* No concurrent radiotherapy

  * Localized radiotherapy to a non-indicator lesion for pain relief allowed provided all other methods of pain control are ineffective

Surgery

* At least 4 weeks since prior major surgery and recovered

Other

* At least 4 weeks since prior myelosuppressive therapy
* At least 4 weeks since prior investigational drugs
* No other concurrent investigational drugs
* No other concurrent anticancer cytotoxic therapy

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-04; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pagan, Study Chair — Daiichi Sankyo
Locations (6):
- United States (5):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
- Veterans Affairs Medical Center - San Juan, San Juan, Puerto Rico

REFERENCES:
- [Result] Patel S, Keohan ML, Saif MW, Rushing D, Baez L, Feit K, DeJager R, Anderson S. Phase II study of intravenous TZT-1027 in patients with advanced or metastatic soft-tissue sarcomas with prior exposure to anthracycline-based chemotherapy. Cancer. 2006 Dec 15;107(12):2881-7. doi: 10.1002/cncr.22334. PMID 17109446